CLINICAL TRIAL: NCT07152678
Title: A Phase II Study of High-Dose-Rate Esophageal Brachytherapy After External Beam Radiotherapy and Nivolumab in Patients With Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Brachytherapy With Radiotherapy and Immunotherapy: Guided HDR Trial in Esophageal Squamous Cell Carcinoma
Acronym: BRIGHT-ESCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202505130MIND
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-07

CONDITIONS: Esophageal Cancer; Esophageal Squamous Cell Carcinoma
Keywords: Esophageal squamous cell carcinoma; Brachytherapy; Immune checkpoint inhibitor; Nivolumab; Radiotherapy; Locoregional control
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — Nivolumab; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Add-on of intraluminal brachytherapy with applicator (Experimental): Brachytherapy protocol starts within 3 weeks after first cycle of immunotherapy administered (This is "week 1"). High-dose-rate (HDR) 5-6 Gy per fraction is delivered to GTV of esophageal tumor(s), second treatment if applicable will be finished within 2 weeks after the first fraction, a total of 5-12 Gy in 1-2 fractions will be delivered. GTV coverage D90 should equal 100% of prescription. It is NOT allowed to give concurrent chemotherapy on the days of HDR brachytherapy.
  Interventions: Drug: Nivolumab (240 mg); Radiation: Brachytherapy

INTERVENTIONS:
Drug: Nivolumab (240 mg) — After the first cycle of nivolumab administered in the screening phase (1st cycle), nivolumab in the study phase was administered intravenously over 30 minutes at a dose of 240 mg every 2 weeks for at least 2 doses, with 1 cycle after to first brachytherapy (2nd cycle), and 1 more cycle after to second brachytherapy (3rd cycle) if feasible. (each cycle was 2 weeks), until disease progression assessed by the investigator per RECIST version 1.1, or unacceptable toxicity.
Radiation: Brachytherapy — Brachytherapy protocol starts within 3 weeks after first cycle of nivolumab was administered. After brachytherapy applicator placement, CT simulation scan(s) with dummy source in place will be done for further planning procedure, including adjustment of the applicator and 3D treatment planning. High-dose-rate (HDR) 5-Gy per fraction is delivered to the gross tumor volume (GTV) of esophageal tumor(s), second treatment if applicable will be finished within 2 weeks after the first fraction, a total of 5-12 Gy in 1-2 fractions will be delivered. GTV coverage D90 should equal 100% of prescription. Efforts should be made to spare the adjacent normal organ and to avoid hot spot on normal esophageal mucosa. It is NOT allowed to give concurrent chemotherapy on the days of HDR brachytherapy.

SUMMARY:
The goal of this clinical trial is to learn if adding high-dose-rate (HDR) brachytherapy can improve outcomes in patients with locally advanced esophageal squamous cell carcinoma (ESCC) who have already received external beam radiotherapy (EBRT), chemotherapy, and the immune therapy drug nivolumab.

The main questions it aims to answer are:

* Does HDR brachytherapy reduce the chance of the cancer coming back in the esophagus or nearby areas within 12 months?
* What side effects or safety issues occur when HDR brachytherapy is given after EBRT, chemotherapy, and nivolumab?

Participants will:

* Receive 1-2 sessions of HDR brachytherapy delivered through a thin tube placed inside the esophagus, within three weeks after starting nivolumab.
* Continue nivolumab and be monitored with regular follow-up visits, imaging tests, and blood samples to check treatment response and safety.

DETAILED DESCRIPTION:
This is a single-arm, phase II clinical trial designed to evaluate the efficacy and safety of high-dose-rate (HDR) esophageal brachytherapy in combination with external beam radiotherapy (EBRT), chemotherapy, and immune checkpoint inhibition with nivolumab in patients with locally advanced esophageal squamous cell carcinoma (ESCC).

Eligible patients include those with stage III-IVB ESCC who have previously received EBRT with concurrent platinum-fluoropyrimidine chemotherapy and who have initiated nivolumab therapy. HDR brachytherapy (5-12 Gy in 1-2 fractions) will be administered within three weeks following the start of nivolumab.

The primary endpoint is the 12-month cumulative incidence of locoregional failure. Secondary endpoints include overall survival, progression-free survival, overall response rate, disease control rate, safety and tolerability, tube-dependence-free survival, tumor-infiltrating lymphocyte density, and circulating tumor DNA dynamics.

The rationale for this trial is that HDR brachytherapy offers precise dose escalation directly to the esophageal tumor, which may improve locoregional control beyond EBRT alone. In addition, the combination of localized high-dose irradiation with systemic immune checkpoint inhibition has the potential to enhance antitumor immunity, thereby improving clinical outcomes in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-85 years, with ECOG performance 0-2.
* Locally-advanced esophageal squamous cell carcinoma with clinical stage III, IVA with biopsy proven.
* Prior treatment with EBRT (40-50.4 Gy in 20-28 fractions) and platinum + fluoropyrimidine chemotherapy, with residual or progressive disease, and deemed inoperable or unable to undergo surgery.
* No prior exposure to ICIs and had received first cycle of nivolumab after CCRT.
* Biopsy proven with PD-L1 [tumor cell (TC) ≥ 1%]
* Required at least one measurable or non-measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1.
* Patients with limited stage IVB disease (e.g., non-visceral lymph node metastasis) may be enrolled if the primary tumor is locally dominant and suitable for brachytherapy, based on investigator's discretion.

Exclusion Criteria:

* Current or past history of severe hypersensitivity to any other antibody products.
* Patients with any metastasis in the brain or meninx that is symptomatic or requires treatment.
* Patients with active, known or suspected autoimmune disease
* Stenosis of esophageal lumen that cannot performed brachytherapy
* Involvement of tracheal mucosa or bronchial mucosa.
* The distribution of the lesions of interest exceeds 10 cm range.
* The patient is participating in other interventional clinical trials associated with immunotherapy.
* The patient is scheduled to undergo esophagostomy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of locoregional failure at 12 months | 12 months from initiation of HDR brachytherapy
  The proportion of patients who develop tumor recurrence or persistence in the esophagus or regional lymph nodes, as assessed by central review using endoscopy, CT and/or PET according to RECIST v1.1 and iRECIST criteria.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 24 months
  Percentage of patients achieving complete response or partial response as best overall response, assessed by investigators per RECIST v1.1 and iRECIST.
Overall Survival (OS) | Up to 24 months
  Time from enrollment to death from any cause.
Progression-Free Survival (PFS) | Up to 24 months
  Time from enrollment to first documented tumor progression or death, whichever occurs first.
Disease Control Rate (DCR) | Up to 24 months
  Percentage of patients achieving complete response, partial response, or stable disease, as best overall response per RECIST v1.1/iRECIST.
Duration of Response (DoR) | Up to 24 months
  Time from the first documentation of complete or partial response to the first documented tumor progression or death.
Cumulative incidence of distant failure | Up to 24 months
  Proportion of patients developing new distant metastases over the study period, accounting for competing risks.
Safety and tolerability | From first study treatment through 90 days after last dose and up to 24 months for late effect
  Incidence and severity of adverse events (AEs), serious adverse events (SAEs), and immune-related adverse events, graded according to CTCAE v5.0.
Tube-dependence-free survival | Up to 24 months
  Proportion of patients who remain alive without requiring feeding tube support (e.g., nasogastric or jejunostomy tube) for nutrition.
Circulating tumor DNA (ctDNA) dynamics | Baseline and up to 24 months
  Change in ctDNA levels measured at baseline and during follow-up as an indicator of treatment response and disease progression.
Tumor-infiltrating lymphocyte (TIL) density | Baseline to up to 12 weeks after HDR brachytherapy
  Change in tumor-infiltrating lymphocyte density in tumor biopsy samples collected before and after HDR brachytherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Ting Liu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital Yunlin Branch, Huwei, Yunlin County, Taiwan